CLINICAL TRIAL: NCT00003690
Title: Phase I Study of Flavopiridol in Combination With Cisplatin in Patients With Advanced Malignancies
Brief Title: Flavopiridol Plus Cisplatin or Carboplatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Keith C. Bible, M.D., Ph.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000066793; U01CA069912 (NIH); P30CA015083 (NIH); 950101 (Other: Mayo Clinic Cancer Center); 276-97 (Other: Mayo Clinic IRB)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer; Melanoma (Skin); Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV breast cancer; recurrent breast cancer; stage IV prostate cancer; recurrent prostate cancer; stage IV melanoma; recurrent melanoma; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Breast Neoplasms; Melanoma; Prostatic Neoplasms | interventions — alvocidib; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: alvocidib
Drug: carboplatin
Drug: cisplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of flavopiridol plus cisplatin or carboplatin in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of flavopiridol and cisplatin in patients with advanced solid tumors. (Part 1)
* Determine the MTD of carboplatin when combined with flavopiridol in another group of patients with advanced solid tumors. (Part 2)
* Determine the toxic effects of these regimens in this patient population.
* Determine the objective clinical response in patients treated with this regimen.
* Determine the pharmacokinetics of these regimens in this patient population.

OUTLINE: This is a dose-escalation study of flavopiridol and cisplatin (part 1), followed by a dose-escalation study of carboplatin (part 2).

* Part 1: Patients receive flavopiridol IV over 24 hours. Two weeks later, patients receive cisplatin IV over 2 hours immediately followed by flavopiridol IV over 24 hours. Treatment with cisplatin/flavopiridol continues every 3 weeks in the absence of unacceptable toxicity or disease progression.

Sequential dose escalation of flavopiridol is followed by sequential dose escalation of cisplatin. Cohorts of 3-6 patients receive escalating doses of flavopiridol and then cisplatin until the maximum tolerated dose (MTD) of the combination is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

* Part 2: Additional patients are accrued for part 2. Those patients receive carboplatin IV over 30 minutes immediately followed by flavopiridol IV over 24 hours. Treatment continues every 3 weeks in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of carboplatin until the MTD is determined. The MTD is defined as in part 1.

PROJECTED ACCRUAL: Approximately 36-48 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable advanced solid tumor for which no standard therapy exists that is potentially curative or definitely capable of extending life expectancy

  * Biopsy confirmation of recurrent tumors required, unless sole site of disease is inaccessible bony and/or pulmonary metastases
* Eligible solid tumors include, but not are limited to, prostate cancer, breast cancer, or melanoma
* No lymphoma
* No CNS metastases

  * Patients with primary brain tumors are eligible if they are not receiving antiepileptic medication(s) but are receiving stable doses of corticosteroids
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* See Disease Characteristics
* At least 12 weeks

Hematopoietic:

* WBC at least 3,500/mm^3
* Absolute neutrophil count at least 1,700/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic:

* Bilirubin within upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No history of angina

Neurologic:

* No grade 2 or greater peripheral neuropathy
* No seizure disorder

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 4 weeks since prior immunotherapy
* More than 4 weeks since prior biologic therapy
* No concurrent immunotherapy

Chemotherapy:

* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosoureas) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 1998-12; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith C. Bible, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States